CLINICAL TRIAL: NCT02263612
Title: Late Mesh Complications After 3258 Incisional Hernia Operations
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: DK_02
Record Dates: First submitted 2014-09-20; First posted 2014-10-13 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Incisional Hernia
Keywords: Incisional Hernia; Complications; Long-term
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Danish Hernia Database: Patients registered in the Danish Ventral Hernia Database during January 1st 2007 to december 31st 2010

SUMMARY:
The Danish Hernia Database (DHD) registers 37 different perioperative parameters. The aim of present study is to use large-scale data from DHD to uncover risk factors for long-term (30 days postoperative and later) readmission, reoperation, death and reoperation for recurrence after incisional hernia repair with use of a synthetic mesh.

DETAILED DESCRIPTION:
All principal incisional hernias registered in the Danish Hernia Database are included in the study. The included patients have been followed for more than 4 years in order to identify correlation between technical aspects of the hernia repair and postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Incisional Hernia Repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All incisional hernia repairs registered in tha Danish National Hernia Database from January 1st 2007 to December 31st 2010
Sampling Method: Non-Probability Sample
Enrollment: 3258 (Actual)
Dates: Start 2007-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Reoperation | Up to 7 years
  Riskfactors for reoperation (any procedure) more than 30 days after incisional hernia repair

SECONDARY OUTCOMES:
Readmission | Up to 7 years
  Riskfactors for readmission later than 30 days after incisional hernia repair

OTHER OUTCOMES:
Death | Up to 7 years
  Riskfactors for death later than 30 days after incisional hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Dunja Kokotovic, MS, Principal Investigator — dept. of surgery, Køge University Hospital
Locations (1):
- Køge Sygehus, Køge, Denmark